CLINICAL TRIAL: NCT01861769
Title: Implementation of Evidence-based Psychotherapy for PTSD: An Empirical Investigation of Post-workshop Consultation in Treatment Fidelity and Patient Outcomes
Brief Title: Implementation of Evidence-based Psychotherapy for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Candice Monson, Professor & Director of Clinical Training, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIHR 2011-03-01
Record Dates: First submitted 2013-05-15; First posted 2013-05-24 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Cognitive Processing Therapy; Consultation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Technology-enhanced Teleconsultation (Experimental): Technology-enhanced Group Tele-consultation. This consultation method requires that participants be prepared to review and receive feedback on audiorecorded CPT sessions in a group format. The CPT expert randomly selects two clinician sessions each week that have been audiorecorded to use for feedback and discussion in group teleconference based on procedures used in previous training initiatives (Stirman, Bhar, et al., 2010). Five- to twenty-minute segments of the two sessions will be shared within the group consultation. The CPT expert will provide feedback on the sessions with an emphasis on review of key learning points. These consultation group sessions will be facilitated with collaborative meeting software that includes audio file uploading.
  Interventions: Other: Technology-enhanced Teleconsultation
- Standard Teleconsultation (Experimental): Standard Tele-consultation Group. The CPT expert will randomly select clinicians for case presentation each week. Each clinician will be responsible for verbally presenting on their CPT cases throughout the 6-month period of consultation course. No audiorecorded content will be reviewed within the calls. All other procedures used in the above condition will be used here.
  Interventions: Other: Standard Teleconsultation
- No consultation (No Intervention): No Consultation/Fidelity Monitoring Only. Participants assigned to this condition will receive no post-workshop expert consultation, but will be subject to the same audiorecorded session-uploading and client-outcome reporting as the other conditions. This condition allows us to assess the effect of clinicians knowing that their sessions are subject to fidelity assessment.

INTERVENTIONS:
Other: Technology-enhanced Teleconsultation — Technology-enhanced Group Tele-consultation. This consultation method requires that participants be prepared to review and receive feedback on audiorecorded CPT sessions in a group format. The CPT expert randomly selects two clinician sessions each week that have been audiorecorded to use for feedback and discussion in group teleconference based on procedures used in previous training initiatives (Stirman, Bhar, et al., 2010). Five- to twenty-minute segments of the two sessions will be shared within the group consultation. The CPT expert will provide feedback on the sessions with an emphasis on review of key learning points. These consultation group sessions will be facilitated with collaborative meeting software that includes audio file uploading.
  Arms: Technology-enhanced Teleconsultation
Other: Standard Teleconsultation — Standard Tele-consultation Group. The CPT expert will randomly select clinicians for case presentation each week. Each clinician will be responsible for verbally presenting on their CPT cases throughout the 6-month period of consultation course. No audiorecorded content will be reviewed within the calls. All other procedures used in the above condition will be used here.
  Arms: Standard Teleconsultation

SUMMARY:
Approximately 9% of Canadians will have Posttraumatic Stress Disorder (PTSD) in their lifetime. In the military veteran population, the lifetime prevalence of PTSD has been estimated to be as high as 20%. Numerous research studies have demonstrated that short-term, cognitive-behavioral psychotherapies, such as Cognitive Processing Therapy (CPT), lead to substantial improvements in PTSD symptoms. However, research suggests that a minority of clinicians provide these therapies in clinical settings. The transfer of this research knowledge into clinical settings remains one of the largest hurdles to improving the health of Canadians with PTSD.

It is well established that attending a 2-day workshop on these therapies alone is insufficient to promote adequate knowledge transfer and sustained skillful use. The current study aims to contrast whether two forms of post-workshop support (6-month duration), with different levels of expert oversight, will result in superior levels of clinician skill and patient outcomes versus no formal post-workshop support. The three forms of post-workshop support are 1) technology-enhanced group tele-consultation 2) standard group tele-consultation 3) no tele consultation. The primary and secondary outcomes will be the assessment of the clinicians' competence in CPT and patient symptoms,respectively. This study will inform how best to transfer evidence based therapy outcomes to the clinical milieu to attain comparable outcomes as those observed in research.

The investigators' hypotheses are as follows: Hypothesis 1:The technology enhanced group tele-consultation condition will evidence the highest levels of fidelity, the standard group tele-consultation condition will evidence intermediate levels of fidelity, and the no-consultation/fidelity monitoring only condition will evidence the lowest fidelity. Hypothesis 2: Fidelity to the CPT protocol, irrespective of consultation condition, will be positively associated with improved client outcomes. Hypothesis 3: Organizational context variables, such as the organizational climate and readiness for change, will influence the uptake of CPT skills, as well as the extent to which these skills are utilized in practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinician participants (n=120) recruited for this study will either be Operation Stress Injury (OSI) network clinicians, Operational Trauma and Stress Support Centre (OTSSC) network clinicians or community-based clinicians who treat military-related PTSD.
* Both male and female clinician participants will be recruited;
* Clinician participants will be greater than 18 years.

Mental health clinicians from the clinics and private practitioners will be eligible to participate in the study if they:

1. attend the CPT workshop;
2. are employees of an OSI or OTSSC clinic, are registered VAC clinicians, or are in private practice treating individuals with military-related PTSD;
3. currently provide psychotherapy to military soldiers or veterans with PTSD;
4. consent to be randomized to one of the three study conditions; and,
5. are willing to solicit patient participation.

Eligible patient participants are:

1. client of the clinician participant, who has a diagnosis of PTSD, as determined by clinician independent assessment, and total PCL score equal or greater to 45; and
2. willing to consent to have their sessions audiorecorded and listened to by a fidelity rater and potentially other clinicians teaching and learning CPT. Patients are permitted to continue other psychotherapeutic interventions if not specifically focused on treating PTSD symptoms. Patient participants must be over the age of 18.

Exclusion Criteria:

Ineligible patients will include those not eligible for CPT based on the state of research evidence, including those with:

1. current uncontrolled psychotic or bipolar disorder;
2. unremitted substance dependence diagnosis (substance abuse allowed);
3. current imminent suicidality or homicidality that requires imminent attention; and
4. significant cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Cognitive Processing Therapy Fidelity Ratings | Clinician-participants' CPT session audio tapes from the 6 month study period will be assessed at the 6 month time point.
  Cognitive Processing Therapy (CPT) sessions will be rated by trained CPT Fidelity raters for fidelity to the CPT protocol.

SECONDARY OUTCOMES:
PTSD Checklist (PCL-S) | At baseline, approximately once per week for approximately 12 weeks, and once at 3 month follow up
  The PCL is a 17-item self-report measure of the 17 DSM-IV symptoms of PTSD.
SF-12 Health Survey | At baseline, approximately once every 2 weeks for approximately 12 weeks, and once at 3 month follow up
  An even shorter - 1-page, 2-minute - survey form has been shown to yield summary physical and mental health outcome scores that are interchangeable with those from the SF-36® in both general and specific populations. This short-form - the SF-12® - which was published in early 1995 is already one of the most widely used surveys.
Outcomes Questionnaire 45 (OQ-45) | At baseline, approximately once per week for 12 weeks, and once at 3 month follow up
  The OQ®-45.2 measures functioning in 3 domains: Symptom distress (heavily loaded for depression and anxiety), Interpersonal functioning, and Social Role. It enables the clinician to assess functional level and change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Candice Monson, Ph D, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Edmonton Operational Stress Injury Clinic, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Wiltsey Stirman S, Shields N, Deloriea J, Landy MS, Belus JM, Maslej MM, Monson CM. A randomized controlled dismantling trial of post-workshop consultation strategies to increase effectiveness and fidelity to an evidence-based psychotherapy for Posttraumatic Stress Disorder. Implement Sci. 2013 Aug 1;8:82. doi: 10.1186/1748-5908-8-82. PMID 23902798